CLINICAL TRIAL: NCT04125849
Title: Mediastinoscopy-assisted Transhiatal Esophagectomy (MATHE) Versus Thoraco-laparoscopic Esophagectomy (TLE) for Esophageal Cancer: a Multicenter Randomized Controlled Trial
Brief Title: Mediastinoscopy-assisted Transhiatal Esophagectomy Versus Thoraco-laparoscopic Esophagectomy for Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Peking University Cancer Hospital & Institute (Other); Hubei Cancer Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Quanzhou First Hospital (Other); The People's Hospital of Gaozhou (Other); The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Mu Juwei, MD，PHD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC201819B69
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Esophageal Neoplasms
Keywords: Mediastinoscopy-assisted transhiatal esophagectomy (MATHE); Thoraco-laparoscopic esophagectomy (TLE)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoraco-laparoscopic esophagectomy (Active Comparator): Treated by thoraco-laparoscopic esophagectomy in the centers with enough experience in esophageal resection and the volume ≧80 cases each year.
  Interventions: Procedure: Thoraco-laparoscopic esophagectomy
- Mediastinoscopy-assisted transhiatal esophagectomy (Active Comparator): Treated by mediastinoscopy-assisted transhiatal esophagectomy in the centers with enough experience in esophageal resection and the volume ≧80 cases each year.
  Interventions: Procedure: Mediastinoscopy-assisted transhiatal esophagectomy

INTERVENTIONS:
Procedure: Thoraco-laparoscopic esophagectomy — Thoraco-laparoscopic esophagectomy surgery
  Arms: Thoraco-laparoscopic esophagectomy
Procedure: Mediastinoscopy-assisted transhiatal esophagectomy — Mediastinoscopy-assisted transhiatal esophagectomy surgery
  Arms: Mediastinoscopy-assisted transhiatal esophagectomy

SUMMARY:
Esophageal cancer is one of the major diseases that seriously threatens an individual's health and life. To reduce the incidence of postoperative complications and mortality of esophageal cancer, thoraco-laparoscopic oesophagectomy (TLE) has been recommended by many guidelines since the 2000s. Additionally, with developments in endoscopy technology in recent years, mediastinoscopy-assisted transhiatal esophagectomy (MATHE) has been used in clinical practice. In 2015, the first mediastinoscopy combined with laparoscopic radical esophagectomy was reported systematically by Hitoshi Fujiwara. This surgical procedure has been performed in many centres in China. However, there is no multicentre prospective randomized controlled study that explored the safety, feasibility and short-term clinical efficacy between mediastinoscopy-assisted transhiatal esophagectomy and thoraco-laparoscopic esophagectomy. We aim to evaluate the feasibility and safety of MATHE.

DETAILED DESCRIPTION:
Esophageal resection remains the mainstay of treatment for esophageal cancer patients. Despite improvements in surgical technique and perioperative management, esophagectomy carries considerable operative risk. To reduce the incidence of postoperative complications and mortality of esophageal cancer, the optional of minimally invasive esophagectomy has been recommended by many guidelines since 2000s. In addition, with the development of endoscopy technology in recent years, mediastinoscopy-assisted transhiatal esophagectomy (MATHE) has been used in clinical practices. In 2015, the first mediastinoscopy combined with laparoscopic radical esophagectomy was reported systematically by Hitoshi Fujiwara. This surgical procedure has been performed in many centers of China since then. Compared with MIE, MATHE allows controlled dissection of upper mediastinum and biopsy of mediastinal lymph nodes. No study directly comparing MATHE versus MIE has been reported to date. In this report, we compare MATHE with MIE in terms of surgical feasibility, safety, and survival.We intend to adopt a randomized controlled study method. The study group is mediastinoscopy-assisted transhiatal esophagectomy (MATHE) group, and the control group is thoraco-laparoscopic esophagectomy (TLE) group. This study is expected to provide high-level evidence for the new methods and to provide better treatment options for patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years≤age≤ 80 years;
* Histologically diagnosed with squamous cell carcinoma by endoscopic biopsy, cT1-3N0M0;
* Primary tumour is located in the thoracic oesophagus
* No clinical evidence of distant organ metastasis
* No severe comorbidity, can tolerate anesthesia;
* ECOG PS scores≤2;
* The patients sign informed consents by themselves.

Exclusion Criteria:

* Cervical or abdominal oesophageal carcinoma;
* Previous oesophagectomy, gastrectomy, or mediastinal surgery;
* Current uncontrolled illness such as severe cardiac disease, uncontrollable hypertension or diabetes, or active bacterial infection;
* Unable to tolerate tracheal intubation and general anaesthesia as determined by an anaesthesiologist preoperatively;
* Pregnant or lactating women;
* ECOG PS scores>2;
* Considered unsuitable, such as those who do not agree to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative respiratory complications | 30 days after surgery
  These respiratory complications involve respiratory distress or failure after the operation with continuation of mechanical ventilation, pulmonary atelectasis requiring sputum suction by bronchoscopy, pneumonia requiring specific antibiotics confirmed by thoracic X-ray or CT scan of the thorax and a positive sputum culture, and acute respiratory distress syndrome.

SECONDARY OUTCOMES:
pulmonary function indicators | 30 days after surgery
  pulmonary function indicators
anastomotic fistula | 30 days after surgery
  anastomotic fistula
recurrent laryngeal nerve palsy | recurrent laryngeal nerve palsy
  recurrent laryngeal nerve palsy
DFS | 3 years
  Disease-free survival,DFS
duration of surgery | Intraoperation
  Total operation time
Blood loss | Intraoperation
  blood loss during the surgery
Conversion rate | Intraoperation
  conversion to thoracotomy during surgery
postoperative hospital stay | postoperation
  postoperative hospital stay
postoperative pain score | postoperation
  postoperative pain score
drainage time | postoperation
  drainage time
R0 resection rate | Intraoperation
  R0 resection rate
Lymph node dissection | Intraoperation
  During the surgery, lymph node dissection were performed. The number of removed lymph-nodes were recorded according to the postoperative pathological diagnosis, and the stations of the lymph node were recorded.
Local recurrence | 3 years
  three-year local tumour recurrence or distant metastasis rate after surgery
30-day mortality after surgery | postoperation
  30-day mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Juwei Mu, MD, Principal Investigator — National Cancer Center of China
Locations (1):
- Cancer Hospital of Chinese Academy of Medical Sciences Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No